CLINICAL TRIAL: NCT05129761
Title: Clinical Response of Syrup Hydryllin® in Pakistani Subjects With Cough in Routine Practice
Acronym: HYD-EFFECT
Status: Completed | Type: Observational
Sponsor: The Searle Company Limited Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCL_HYD-EFFECT-001
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cough
Keywords: Cough management, Cough syrup, Quality of Life
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- • Patient with a clinical history of cough: Syrup Hydryllin ( Syrup Hydryllin & Hydryllin Sugar-Free (Diphenhydramine, Ammonium Chloride, Menthol, Aminophylline) and Syrup Hydryllin DM (Dextromethorphan & Diphenhydramine) in the symptomatic management of cough in routine practice by physicians. Subjects will be observed for overall safety and effectiveness of study drug from visit 1 (baseline visit, screening, and start of treatment), to visit 2 (Week 1-2, end of treatment) in the routine practice.
  Interventions: Drug: Syrup Hydryllin

INTERVENTIONS:
Drug: Syrup Hydryllin — ( Syrup Hydryllin & Hydryllin Sugar-Free (Diphenhydramine, Ammonium Chloride, Menthol, Aminophylline) and Syrup Hydryllin DM (Dextromethorphan & Diphenhydramine)

SUMMARY:
A cough is one of the most common medical complaints accounting for as many as 30 million clinical visits per year. It is the single most prevalent symptom on presentation to a physician's office. Up to 40% of these complaints result in a referral to a pulmonologist. Although, the cough is an essential defense mechanism, still, chronic cough may cause significant morbidity and substantially affect the quality of life and psychosocial wellbeing.

DETAILED DESCRIPTION:
Globally, the prevalence of acute cough is 9 to 64%, whereas chronic cough is >10% in most countries or regions, ranging from 7.2%-33%. In Pakistan, a few studies have examined chronic cough resulting from specific occupations, such as those involving brick kilns, textile work, or gem cutting. Additionally, 15.8% of subjects in a periurban area of Karachi City, Pakistan with cough lasting ≥ 2 weeks were found to have pulmonary TB. Overall, to estimate the prevalence and incidence of different coughs, there is no data available based on the local population, and the data assessing the quality of life of patients with different coughs is not available. Locally, few studies were conducted on cough syrups with a small sample size. However, no real data is available for the symptomatic management of cough about the patient's quality of life related to different coughs. The current study is designed to assess the response of different strengths of Syrup Hydryllin ( Syrup Hydryllin & Hydryllin Sugar-Free (Diphenhydramine, Ammonium Chloride, Menthol, Aminophylline) and Syrup Hydryllin DM (Dextromethorphan & Diphenhydramine) in the symptomatic management of cough in routine practice by physicians. The study's main objective is to assess the quality of life of the subjects suffering from the different types of cough.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical history of cough.
* Patients aged ≥12 and ≤70 years inclusive of either sex.
* The patient will be screened for COVID-19
* The patient will be prescribed the study drug following an approved package insert
* Written informed consent before participation in study-specific procedures

Exclusion Criteria:

* Known hypersensitivity to Hydryllin product, the metabolites, or formulation excipients.
* Covid Patients with moderate and severe condition requires hospitalization or/and associated with the complications.
* Patients who have a contra-indication (refer to the Syrup Hydryllin prescribing information).
* Pregnant (assessed on LMP)
* Breastfeeding women (assessed on interview).

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population including patients of either sex between ≥12 and ≤70 years, suffering from cough (acute, subacute, and chronic), will be enrolled in the study in the random order. The random number will be marked using a random number table.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
• To assess the effectiveness of Syrup Hydryllin from baseline to 2 weeks - | 4 Months
  The effectiveness assesses by Leicester Cough Questionnaire (QoL questionnaire), The LCQ scale from 1-7, 1 is all the time and 7 is none of the time. The total score is 19 whereas 8 for Physical, 7 for Psychological and 4 for Social.

SECONDARY OUTCOMES:
• To assess the overall safety of different strengths of Syrup Hydryllin in the cases presenting with different types of cough. | 4 Months
  The safety will be monitored from the first dose of HYDRYLLIN. The participants with treatment-related adverse events will be reported on Searle AE designed form.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Sarwar, Study Director — The Searle Company Limited
Locations (1):
- The Searle Company Limited, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No